CLINICAL TRIAL: NCT05440279
Title: Effects of an Early Combination of Automated Electronic and Telemedical Support on the Therapeutic Results of CPAP and APAP Patients and as a Supplement to (Tele-) Medical Care
Brief Title: Effects of Telemedical Support on Therapeutic Results of CPAP Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Facharztzentrum Sonneberg-Coburg uBAG (Other)
Collaborators: Heinen und Löwenstein GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2947
Record Dates: First submitted 2022-06-15; First posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Obstructive Sleep Apnea; Adherence, Treatment
Keywords: Interventional; randomized; adherence; continuous positive airway pressure; CPAP; telehealth; obstructive sleep apnea; digital patient support; prisma APP
MeSH Terms: conditions — Sleep Apnea, Obstructive; Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: National, monocentric, prospective, randomized and controlled clinical trial with 2 arms.
  Arm 1: Control group - Standard Care (SC) Arm 2: Intervention group - Standard Care (SC) + digital patient support (DPS) tool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (SC) (No Intervention): Treatment in the control group takes place as standard care that includes an education session with a respiratory therapist about OSA and its consequences, proper use and maintenance of the CPAP device and mask, and therapy and study expectations, provision with a fixed or auto CPAP device (prismaSMART/ prismaSOFT, Löwenstein Medical Technology GmbH & Co. KG), a heated humidifier (prismaAQUA, Löwenstein Medical Technology GmbH & Co. KG) if needed, and a fitting interface, the initiation of therapy with anamnesis, diagnosis night, titration night, education, etc., as well as standardized therapy control after 12 weeks.
- Standard Care (SC) + digital patient support (DPS) tool (Active Comparator): Treatment in the intervention group takes place as standard care (please see description of arm 1 - control group) and electronic therapy support in addition. The electronic therapy support consists of:
  1. Emails to patients with personalized, automated feedback on their therapy (derived from device data received via modem or data entered by the patient via electronic questionnaire),
  2. electronic questionnaires (web-based) on possible problems during therapy, personal adherence goals and subjective therapy success,
  3. possibility to set personal adherence goals every week,
  4. links to explanations and videos on therapy and the handling of therapy equipment and accessories,
  5. provision of data for the trial center in the event of contact by the patient, as well as for routine therapy monitoring.
  Interventions: Device: digital patient support

INTERVENTIONS:
Device: digital patient support — Intervention takes place through a regular electronic therapy support in addition to standard care that is defined as follows:
  Emails to patients with personalized, automated feedback on their therapy (derived from device data received via modem or data entered by the patient via electronic questionnaire),
  1. electronic questionnaires (web-based) on possible problems during therapy and subjective therapy success,
  2. possibility to set personal adherence goals every week,
  3. links to explanations and videos on therapy and the handling of therapy equipment and accessories,
  4. provision of data for the trial center in the event of contact by the patient, as well as for routine therapy monitoring.
  Arms: Standard Care (SC) + digital patient support (DPS) tool

SUMMARY:
Obstructive sleep apnea (OSA) is a type of sleep-related breathing disorders that is characterized by a sleep-related constriction (obstruction) of the upper airways. The treatment with continuous application of positive airway pressure (CPAP) via respiratory mask forms the therapeutical standard of OSA. The autoCPAP (automatic positive airway pressure: APAP) therapy is an additional treatment option for patients with more unstable conditions (e.g. due to sleep position) which is characterized by a dynamic adaption of the applied airway pressure according to patients therapeutical needs. Device usage time and therapy adherence are crucial for treatment success.

The purpose of this study is to assess the effect of a digital patient support (DPS) tool, complementary to standard care on continuous and automatic positive airway pressure (CPAP, APAP) adherence and daytime sleepiness after 12 weeks in patients diagnosed with severe obstructive sleep apnea (OSA).

All patients with apnea-hypopnea index (AHI) ≥ 30 per hour are prospectively included and randomized to receive standard care (SC) or standard care with personalized DPS via prisma APP prototype version (SC+DPS). In both arms, initiation of therapy and standardized therapy control after 12 weeks is carried out identically. Patients in the SC+DPS arm received additionally automated feedback on their therapy and motivational messages, as well as therapy recommendations.

DETAILED DESCRIPTION:
Clinical Picture From the epidemiological view obstructive sleep apnea (OSA) is the most common type of sleep-related breathing disorders (SRBD). OSA is characterized by a sleep-related constriction (obstruction) of the upper airways that in adulthood is often caused by a neuromuscular related impairment of the pharyngeal tone. OSA is linked to many negative health consequences and is associated with a large number of comorbidities.

General treatment As a rule SRBD are treated with appropriate therapy devices that transmit positive airway pressure (PAP) via respiratory masks. In the case of the treatment of obstructive sleep apnea (OSA) therapeutical standard is formed by application of continuous positive airway pressure (CPAP). CPAP therapy devices provide a stable positive airway pressure during sleep to prevent the upper airway obstructions. The determination of the essential airway pressure that keeps airways open takes place within the therapy setting night in the sleep laboratory under polysomnographic monitoring. Patients with more unstable pressure needs, e.g. based on position shifts during the night, also qualify for an autoCPAP (APAP) therapy. APAP therapy devices adapt the applied airway pressure dynamically within defined ranges according to patients' therapeutical needs. Therapy success is essentially defined by average device usage time and patients' long-term therapy adherence which in term is affected by a broad variety of factors. The identification of these factors therefore lead to the development of different treatment strategies to improve patients' therapy adherence.

Usual therapeutical process Patients with suspected OSA are surveyed according to their symptomatology and receive a sleep medical examination under polygraphical or polysomnographical observation. During the sleep medical examination numerous cardiorespiratory and somnological signals are recorded and evaluated.

As far as the evaluation of the recorded signals leads to the diagnosis of OSA and no indications for another type of PAP therapy are present, the adjustment to CPAP or APAP therapy under polysomnographical observation takes place immediately after diagnosis.

Following this, patients receive an appropriate adjusted CPAP- or APAP therapy device and get introduced in it´s handling to continue therapy by themselves in their home environment.

As part of the nightly home therapy, patients are expected to use the device according to the physicians advice. During the home therapy phase, the device is recording specific data to subsequently allow to draw conclusions about the therapeutic process and the therapy quality. In case of difficulties with therapy and dependent on their causes, patients are admonished to contact the sleep laboratory (regarding general problems with therapy) or the provider (regarding problems with the respiratory mask or device settings).

After a period of about 12 weeks, patients again appear in person in the sleep laboratory as part of the general therapy control. During the therapy control, the home usage data recorded by the therapy device are printed in reportform and the interventions which were implemented between first therapy setting and the therapy control are evaluated.

Finally, the medicating physician evaluates the therapy success within a conversation with the patients. In case of an inadequate outcome, therapy settings may have to be optimized.

Rationale of the study Literature shows that the first days of home therapy are crucial for long-term therapy adherence and that telemetrical support through automatic feedback can have a positive effect on therapy adherence.

However, there is a lack of experience how the effect on therapy outcomes caused by more individualized, automatic feedbacks combined with an appropriate supply of information and motivation over a longer period can be assessed.

This study is intended to investigate if therapy outcomes of CPAP and APAP patients can be further improved by an early intervention in the form of a combination of telemetric and electronic support.

Description of the applied medical device The applied medical device are the CE certified medical devices prismaSOFT/ prismaSMART (Type WM090TD) made by Löwenstein Medical Techology GmbH und Co. KG Hamburg. The applied accessories (especially breathing tubes, masks, humidifier, modems) are CE certified, too.

Devices of the WM090TD type are pressure-controlled, non-invasive, non-lifesupporting therapy devices or treating sleep-related breathing disorders (SRBDs) using a mask. The devices are used on persons weighing 30 kg or more. CPAP mode can be used on persons aged 3 years upwards. The device may only be used on a physician's instructions. (auto)CPAP mode provides positive airway pressure for treating obstructive sleep apnea in patients who breathe spontaneously.

Devices of the WM090TD type are used in clinical facilities and in the domestic environment. In the domestic environment, the devices also ac-company the owner on trips away.

The application of the device as part of this study takes place according to it´s intended use and within it´s indication range.

Procedure and interventions

If an OSA was diagnosed, patients will be asked for study participation and get informed about the rationale of the study. In case of patients informed consent they will be randomized to one of two groups (Standard Care = control group vs. Standard Care + Digital Patient Support Tool = intervention group).

At baseline, all patients receive an education session with a respiratory therapist about OSA and its consequences, proper use and maintenance of the CPAP device and mask, and therapy and study expectations. All patients are provided with a fixed or auto CPAP device (prismaSMART/ prismaSOFT, Löwenstein Medical Technology GmbH & Co. KG), a heated humidifier (prismaAQUA, Löwenstein Medical Technology GmbH & Co. KG) if needed, and a fitting interface. The initiation of therapy with anamnesis, diagnosis night, titration night, education, etc., as well as standardized therapy control after 12 weeks is carried out identically in standard care (SC) and in standard care with personalized digital support via prototype of prisma APP (SC+DPS) group and according to clinical routine.

At the beginning and with completion of the study every participant is surveyed about his daytime sleepiness applying the standardized questionnaire "Epworth Sleepiness Scale (ESS)".

With completion of the study, each patient furthermore assesses his satisfaction with the CPAP therapy in general and with focus on therapy instructions and support. For this purpose, they rate 8 questions on a scale of 0-4, with a 4 being the best rating (0: strongly disagree, 1: barely disagree, 2: partly agree, 3: mostly agree, 4: strongly agree).

The intervention (SC+DPS) group receives electronic therapy support in addition to standard care. The electronic therapy support consists of:

1. Emails to patients with personalized, automated feedback on their therapy (derived from device data received via modem or data entered by the patient via electronic questionnaire),
2. electronic questionnaires (web-based) on possible problems during therapy and subjective therapy success,
3. possibility to set personal adherence goals every week,
4. links to explanations and videos on therapy and the handling of therapy equipment and accessories,
5. provision of data for the trial center in the event of contact by the patient, as well as for routine therapy monitoring.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80 years
* CPAP-naïve
* confirmed severe OSA (AHI >30/h), diagnosis based on polysomnography (PSG) (MiniScreen PRO with Software MiniscreenViewer, Dr. Fenyves & Gut, Rangendingen, Germany)
* written informed consent to participate in the study, including a data protection statement.

Exclusion Criteria:

* presence of a contraindication to PAP therapy
* participation in another study influencing automated electronic support
* lack of possibility to receive emails or use electronic means of communication
* lack of patient consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Daytime sleepiness (ESS Score) | Baseline and after 12 weeks (Diagnosis/ baseline to therapy control)
  Significant change in daytime sleepiness of CPAP/ APAP patients with standard care plus support of a digital patient support (DPS) tool versus patients with standard care without support of a digital patient support (DPS) tool from baseline at therapy control after 12 weeks

SECONDARY OUTCOMES:
Therapy adherence | Within 12 weeks (period between diagnosis/ baseline to therapy control)
  evaluated by average device usage time in minutes per day and percentual amount of days with an average usage time > 4 hours
Therapy efficacy | Within 12 weeks (period between diagnosis/ baseline to therapy control)
  evaluated by Apnea Hypopnea Index (AHI), obstructive Apnea Hypopnea Index (oAHI), central Apnea Hypopnea Index (cAHI), snoring during diagnosis, polygrahpic therapy control and therapy data stored by therapy device, as well as mask leakage and deep sleep according to therapy data stored by therapy device
type and frequency of usage of device comfort features | Within 12 weeks (period between diagnosis/ baseline to therapy control)
  evaluated by number of types and frequency of device comfort features usage
satisfaction with therapy and care according to standardized survey | up to 12 weeks
  evaluated by survey scores
Investigation of progress of therapy adherence, therapy efficacy and side effects in the intervention group | Within 12 weeks (period between diagnosis/ baseline to therapy control)
  evaluated by observation of the corresponding parameters during duration of study per patient
Investigation of frequency of usage of the DPS (Digital Patient Support) tool in the intervention group | Within 12 weeks (period between diagnosis/ baseline to therapy control)
  evaluated by frequency of DPS tool usage
Investigation of type of usage of the DPS (Digital Patient Support) tool in the intervention group | Within 12 weeks (period between diagnosis/ baseline to therapy control)
  evaluated by number of types of DPS tool usage
Correlation between secondary variables and primary variable to investigate the impact of secondary variables on the primary outcome | up to 12 weeks
  evaluated by descriptive analysis of the corresponding parameters
Investigation of the drop out rate, especially impact of therapy break-off | up to 12 weeks
  evaltuated by number of drop outs due to therapy break-off

CONTACTS AND LOCATIONS:
Overall Officials: Christian Franke, Dr.med., Principal Investigator — Facharztzentrum Sonneberg
Locations (1):
- Facharztzentrum Coburg Sonneberg, Sonneberg, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antic NA, Catcheside P, Buchan C, Hensley M, Naughton MT, Rowland S, Williamson B, Windler S, McEvoy RD. The effect of CPAP in normalizing daytime sleepiness, quality of life, and neurocognitive function in patients with moderate to severe OSA. Sleep. 2011 Jan 1;34(1):111-9. doi: 10.1093/sleep/34.1.111. PMID 21203366
- [Background] Budhiraja R, Parthasarathy S, Drake CL, Roth T, Sharief I, Budhiraja P, Saunders V, Hudgel DW. Early CPAP use identifies subsequent adherence to CPAP therapy. Sleep. 2007 Mar;30(3):320-4. PMID 17425228
- [Background] Hwang D, Chang JW, Benjafield AV, Crocker ME, Kelly C, Becker KA, Kim JB, Woodrum RR, Liang J, Derose SF. Effect of Telemedicine Education and Telemonitoring on Continuous Positive Airway Pressure Adherence. The Tele-OSA Randomized Trial. Am J Respir Crit Care Med. 2018 Jan 1;197(1):117-126. doi: 10.1164/rccm.201703-0582OC. PMID 28858567
- [Background] Kushida CA, Littner MR, Hirshkowitz M, Morgenthaler TI, Alessi CA, Bailey D, Boehlecke B, Brown TM, Coleman J Jr, Friedman L, Kapen S, Kapur VK, Kramer M, Lee-Chiong T, Owens J, Pancer JP, Swick TJ, Wise MS; American Academy of Sleep Medicine. Practice parameters for the use of continuous and bilevel positive airway pressure devices to treat adult patients with sleep-related breathing disorders. Sleep. 2006 Mar;29(3):375-80. doi: 10.1093/sleep/29.3.375. PMID 16553024
- [Background] Lewis KE, Seale L, Bartle IE, Watkins AJ, Ebden P. Early predictors of CPAP use for the treatment of obstructive sleep apnea. Sleep. 2004 Feb 1;27(1):134-8. doi: 10.1093/sleep/27.1.134. PMID 14998250
- [Background] Sawyer AM, Gooneratne NS, Marcus CL, Ofer D, Richards KC, Weaver TE. A systematic review of CPAP adherence across age groups: clinical and empiric insights for developing CPAP adherence interventions. Sleep Med Rev. 2011 Dec;15(6):343-56. doi: 10.1016/j.smrv.2011.01.003. Epub 2011 Jun 8. PMID 21652236
- [Background] Shoib, S., Malik, J. A., Masoodi, S. R., & Rashid, A. (2018). Screening for comorbidities in obstructive sleep apnea. Journal of Clinical and Diagnostic Research, 12(1), VC01-VC03. https://doi.org/10.7860/JCDR/2018/27635.11071
- [Background] Weaver TE, Maislin G, Dinges DF, Bloxham T, George CF, Greenberg H, Kader G, Mahowald M, Younger J, Pack AI. Relationship between hours of CPAP use and achieving normal levels of sleepiness and daily functioning. Sleep. 2007 Jun;30(6):711-9. doi: 10.1093/sleep/30.6.711. PMID 17580592
- [Background] Duran J, Esnaola S, Rubio R, Iztueta A. Obstructive sleep apnea-hypopnea and related clinical features in a population-based sample of subjects aged 30 to 70 yr. Am J Respir Crit Care Med. 2001 Mar;163(3 Pt 1):685-9. doi: 10.1164/ajrccm.163.3.2005065. PMID 11254524
- [Background] Peppard PE, Young T, Barnet JH, Palta M, Hagen EW, Hla KM. Increased prevalence of sleep-disordered breathing in adults. Am J Epidemiol. 2013 May 1;177(9):1006-14. doi: 10.1093/aje/kws342. Epub 2013 Apr 14. PMID 23589584
- [Derived] Franke C, Piezonna F, Schafer R, Grimm A, Loris LM, Schwaibold M. Effect of a digital patient motivation and support tool on CPAP/APAP adherence and daytime sleepiness: a randomized controlled trial. Sleep Biol Rhythms. 2023 Aug 17;22(1):49-63. doi: 10.1007/s41105-023-00479-9. eCollection 2024 Jan. PMID 38469583